CLINICAL TRIAL: NCT05157451
Title: Randomized Prospective Two-Arm Feasibility Trial of Stereotactic Body Radiation Therapy Versus Yttrium-90 Segmentectomy in Inoperable Hepatocellular Carcinoma
Brief Title: Y-90 Versus SBRT for Inoperable HCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not feasible at this time.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: American Society of Clinical Oncology (Other); Medical Research Foundation, Oregon (Other); Oregon Health and Science University (Other); Radiation Oncology Institute (Unknown); Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Nima Nabavizadeh, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: STUDY00022029; NCI-2021-11880 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022029 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma; Stage I Hepatocellular Carcinoma AJCC v8; Stage IA Hepatocellular Carcinoma AJCC v8; Stage IB Hepatocellular Carcinoma AJCC v8; Stage II Hepatocellular Carcinoma AJCC v8; Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Quality of Life; Radiosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (SBRT) (Experimental): Patients undergo SBRT every other day for a total of 5 days over 2 weeks.
  Interventions: Other: Quality of Life; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy
- Arm II (Y-90 radioembolization) (Experimental): Patients receive Y-90 radioembolization via injection on day 1.
  Interventions: Other: Quality of Life; Other: Questionnaire Administration; Procedure: Yttrium-90 Microsphere Radioembolization

INTERVENTIONS:
Other: Quality of Life — Ancillary studies
  Other Names: QOL; quality of life (QoL); Quality-of-Life
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm I (SBRT)
Procedure: Yttrium-90 Microsphere Radioembolization — Given via injection
  Other Names: Yttrium Y 90 Microsphere Therapy; Yttrium-90 Radioembolization
  Arms: Arm II (Y-90 radioembolization)

SUMMARY:
This phase II trial tests whether Y-90 segmentectomy (internal radiation) versus stereotactic body radiation therapy (external radiation) is more optimal in treating inoperable liver cancer. Y-90 segmentectomy consists into very tiny radioactive glass beads that can be injected into the liver through the blood vessels supplying the liver. Stereotactic body radiation therapy uses special equipment to position a patient and deliver external radiation to tumors with high precision. This study many help doctors determine which treatment, Y-90 segmentectomy or SBRT, works better in treating liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine feasibility of trial enrollment (enrollment date).

SECONDARY OBJECTIVE:

I. To assess differences in overall survival, local control, time to intrahepatic progression, time to next treatment, rate of liver transplant, toxicity, and patient reported complications and quality of life.

EXPLORATORY OBJECTIVE:

I. Compare cumulative cost of treatment-related medical care at 13 months.

OUTLINE: Patients will be randomized in 1 of 2 arms.

Arm I: Patients undergo SBRT every other day for a total of 5 days over 2 weeks.

Arm II: Patients receive Y-90 radioembolization via injection on day 1.

After completion of study, patients are followed up at 2, 4, and 12 weeks and then every 3 months for 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age >= 18 years at time of informed consent. Both men and women and members of all races and ethnic groups will be included.
* Patient with non-metastatic hepatocellular carcinoma (HCC) including lesion(s) amenable to definitive therapy with either SBRT or Y-90 segmentectomy, limited to =< 2 liver segments, as agreed upon by the multidisciplinary tumor board consensus.
* Patient not otherwise optimal candidates for resection or thermal ablation, as agreed upon by the multidisciplinary tumor board.
* Have a Child-Pugh criteria (CP) score B7 or better.
* Eastern Clinical Oncology Group (ECOG) performance status =< 1, or Karnofsky performance scale > 70.
* No other prior invasive malignancy is allowed except for the following: adequately treated basal or squamous cell skin cancer, in situ breast or cervical cancer. Stage I or II invasive cancer treated with a curative intent without evidence of disease recurrence for at least five years.

Exclusion Criteria:

* Participant is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, serious or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrollment (enrollment rate) | Up to 4 years
  Determine feasibility of trial enrollment for two therapeutic groups.

SECONDARY OUTCOMES:
Overall survival | Death, adjuvant systemic therapy or liver directed therapy to treated lesion, transplant, lost to follow up, or 13 months post-treatment
Time to progression | Time of radiographic evidence of treated tumor progression as determined by tumor board review, adjuvant systemic therapy or liver directed therapy to treated lesion, transplant, death, or 13 months post-treatment
Time to intrahepatic progression | Time of radiographic intrahepatic progression, adjuvant systemic therapy or liver directed therapy, transplant, death, or 13 months post-treatment
Rate of liver transplant | Time of liver transplant, death, or 13 months post-treatment
Rate of non-classic radiation induced liver disease | Up to 13 months
  Defined as a Child-Pugh criteria >= 2 point increase.
Rate of patient reported outcome-Common Terminology Criteria for Adverse Events | Baseline up to 13 months
Change in patient reported quality of life | Baseline to 13 months
  Measured by Functional Assessment of Cancer Therapy-Hepatobilliary Cancer compared to baseline.
Time to next treatment | Time to next liver directed or non-adjuvant systemic therapy, transplant, or death, assessed up to 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Nima Nabavizadeh, Principal Investigator — OHSU Knight Cancer Institute